CLINICAL TRIAL: NCT03137056
Title: Characterization of Proteins and Forms of Albumin Removal Capacities of the Theranova Membrane by Innovating Proteomic Investigations
Brief Title: Characterization of Removal Capacities of the Theranova Membrane by Proteomic Investigations
Acronym: DIALOMIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 69HCL17_0144
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Dialysis Membrane Reaction
Keywords: Hemodialysis; Membrane; Albumin; Proteomics
MeSH Terms: interventions — Renal Dialysis; Hemodiafiltration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hemodialysis with Theranova (Active Comparator): This arm is represented by the period during which the patients will undergo dialysis with the Theranova membrane.
  Interventions: Device: Hemodialysis with Theranova
- Hemodialysis with FX1000 (Active Comparator): This arm is represented by the period during which the patients will undergo dialysis with the FX1000 membrane.
  Interventions: Device: Hemodialysis with FX1000
- Hemodiafiltration with FX1000 (Active Comparator): This arm is represented by the period during which the patients will undergo dialysis with the FX1000 membrane.
  Interventions: Device: Hemodiafiltration with FX1000

INTERVENTIONS:
Device: Hemodialysis with Theranova — Theranova is a polyarylethersulfone-based hemodialysis membrane manufactured by Baxter International Corp All the dialysis sessions in this arm will be performed with the theranova membrane. This membrane will exclusively be used in hemodialysis.
  Modalities of hemodialysis : Blood flow: 300-400 mL/min; Dialysate flow: 500-800 mL/min
  Arms: Hemodialysis with Theranova
Device: Hemodialysis with FX1000 — FX1000 is a helixone-based membrane manufactured by Fresenius All the dialysis sessions in this arm will be performed with the FX1000 membrane. This membrane will be used in hemodialysis.
  Modalities of hemodialysis: Blood flow: 300-400 mL/min ; Dialysate flow: 500-800 mL/min
  Arms: Hemodialysis with FX1000
Device: Hemodiafiltration with FX1000 — FX1000 is a helixone-based membrane manufactured by Fresenius All the dialysis sessions in this arm will be performed with the FX1000 membrane. This membrane will be used in hemodiafiltration Modalities of hemodialysis: Blood flow: 300-400 mL/min; Dialysate flow: 500-800 mL/min ; post reinjection convection volume of at least 25L.
  Arms: Hemodiafiltration with FX1000

SUMMARY:
Hemodialysis is the major technique of renal suppleance and membrane improvements allow an efficient depuration. During the past fifty years, improving the architecture of the membranes increased constantly the clearance of uremic toxins. Online-hemodiafiltration allowed a potential interest for decreasing morbi-mortality, but this technique is not available in all hemodialysis centers yet. Theranova membrane, by its innovating architecture, could be a valuable option for the enhancement of toxin removal in patients who are not eligible for online-hemodiafiltration techniques. Interestingly, many works pointed adsorptive capacities of dialysis membranes and these observations suggest that adsorption cannot be considered as an epiphenomenon. However, there is a lack of knowledge about the extent of its benefits in hemodialysis. The efficiency of a session of hemodialysis is routinely based on the clearance of only few generic toxins (urea, ß2-microglobulin, myoglobin). The eKT/V formula permitted to link a good depuration of urea with a better survival. EuTox described in a recent review, a large panel of middle molecules considered as uremic toxins. As there are many involved toxins, modern evaluation of hemodialysis efficiency can't be still based on the only description of ß2-microglobulin and urea removals. Inflammation status is routinely measured with blood levels of CRP. However, its accumulation is not leading to a toxicity. Many others inflammatory markers have been linked with morbidity and atherosclerosis, the main cause of mortality in ESRD patients. Obviously, removal of inflammatory markers by different dialyzers needs to be assess concomitantly but single conventional dosages are time-consuming.

A minimal albumin loss is considered as another important factor for a safe hemodialysis. Due to its multiple biological functions, albumin may be one of the most important protein for the maintenance of body homeostasis. Recent works were interested in the potential toxicity of some isoforms of the albumin and especially in chronic kidney disease. Modified forms of albumin have been linked with toxic properties and the removal of modified forms could be beneficial. Furthermore, albumin oxidation can lead to an under-estimation of albumin levels with the routinely used assay. A modern evaluation of the capacities of depuration of dialyzers clearly needs to integrate the evaluation of the clearance and generation of modified forms of albumin and proteins.

Proteomic techniques allow an interesting non-selective integrative approach. This exhaustive view would be particularly adequate for building a snapshot of blood uremic toxins, permeative and adsorptive capacities of each membrane. Due to a high sensitiveness, proteomic techniques can improve dramatically the characterization of the depuration capacities of different hemodialysis membranes considering a large range of uremic toxins especially with middle molecular weight, a large panel of inflammatory markers and modified forms of albumin. Furthermore, proteomic approach can help to build a quasi-exhaustive description of all the proteins removed by a membrane.

This project aims to compare the removal capacities of each membrane on a large range of proteins and forms of albumin (native and modified) with a highly-sensitive LC-MS/MS proteomic approach. We will also build the complete proteome of depuration of each tested membrane.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient on hemodialysis for at least 1 year
* Patient with a functional vascular access permitting at least 300 mL/min of blood flow.

Exclusion Criteria:

* Running infection or other active disease (scheduled surgery, cancer, hospitalisation),
* Catheter as vascular access,
* Recirculation of vascular access over 10%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Comparison of Theranova and FX1000 in high-flux hemodialysis on whole proteome of depuration (qualitative and semi-quantitative description of all the proteins depurated by absorption and convection) | Proteome is evaluated after an 8-weeks session of use of each membrane
  Semi-quantitative analysis is based on the adondance relative of the protein detected on the spectra from the mass spectrometry assay. Quantity will be extrapoled from the level of B2-microglobulin which will be previously assayed in the original samples.

SECONDARY OUTCOMES:
Comparison of Theranova, FX1000 in high-flux hemodialysis and FX1000 in online-hemodiafiltration on differential depuration capacities among albumin isoforms, albumin loss in the dialysate and adsorbed onto the membranes | Isoforms of albumin are evaluated at week 1 and week 8 of use of each membrane and before and after a hemodialysis session during week 1
  Mass excess will be assayed from each amino acid of albumin peptide. This mass excess will be linked with a specific adduct and percentage of presence of each adduct will be calculated.
Comparison of Theranova and FX1000 in high-flux hemodialysis on quantitative removal of protein-bounded toxins and quantitative distribution of inflammatory markers removed by dialysis. | Evaluation after a 8-weeks session of use of each membrane
  Protein-bounded toxins: indoxyl sulfate, p-cresyl sulfate, indole-3 acetic acid - liquid chromatography Inflammatory markers : ET-1, RANTES, MIP-1alpha, MIP-1ß, Eotaxin, MCP-1, Fractalkin, IL-1, IL-2, IL-6, IL-8, IL-10, IL-18, TNF-alpha, C5a, C3a, Factor D, sICAM-1, sVCAM-1, sE-selectin, PAI-1, sFlt-1 - Luminex assay
Comparison of eKT/V of urea and ß2-microglobulin, removal rates and amount in the dialysate of ß2-microglobulin and myoglobin. | Evaluation after a 8-weeks session of use of each membrane
Comparison of serum albumin level after 8 weeks of hemodialysis with (Theranova in hemodialysis, FX1000 in online-hemodiafiltration, FX1000 in hemodialysis) | Evaluation after a 8-weeks session of use of each membrane

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Néphrologie -Hypertension - Hémodialyse, Hôpital Edouard Herriot, Lyon, France